CLINICAL TRIAL: NCT06486168
Title: Incidence of Diaphragmatic Dysfunction After Non-Intubated Video-Assisted Thoracoscopic Surgery.
Acronym: DYNASTY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024-A00912-45
Record Dates: First submitted 2024-06-21; First posted 2024-07-03 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Diaphragmatic Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diaphragmatic Dysfunction evaluation (Experimental)
  Interventions: Procedure: NIVATS

INTERVENTIONS:
Procedure: NIVATS — Non-Intubated Video-Assisted Thoracic Surgery (NIVATS) is the least invasive approach available. It is part of an optimal Enhanced Recovery After Surgery (ERAS) pathway and allows for expanding surgical indications in patients with poor cardio-pulmonary function.

SUMMARY:
The objective of this this single-center prospective longitudinal study is to evaluate the incidence of diaphragmatic dysfunction after non-intubated video-assisted thoracoscopic surgery (NIVATS).

Participant will be evaluated during surgery, 2 hours and 24 hours after surgery.

DETAILED DESCRIPTION:
This is a prospective longitudinal single-center study conducted on patients undergoing non-intubated video-assisted thoracoscopic surgery. The main indications for this surgery are wedge resections, pneumothorax repair, and pleural biopsies (with or without talc pleurodesis) for pleural effusion.

Except for the inclusion visit, each patient will be evaluated twice, 2 and 24 hours after the end of the surgical procedure. The data from each evaluation will be recorded by the physician in the electronic CRF

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or older
* Patient who has read and signed the informed consent form for participation in the study
* Patient undergoing surgery with video-assisted thoracoscopic surgery without intubation

Exclusion Criteria:

* Known or detected diaphragmatic dysfunction before the intervention
* Patient not affiliated with the French social security system
* Patient under legal protection, guardianship, or curatorship
* Patient already enrolled in another therapeutic study protocol (involving medications or non-drug therapies)
* Patient in an exclusion period from a previous clinical study
* Mental deficiency or any other reason that may hinder understanding or strict adherence to the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Diaphragmatic excursion | Hour 24
  The measurement of diaphragmatic excursion at H2 and H24 constitutes the primary evaluation criterion. Diaphragmatic excursion will be measured by ultrasound using a low-frequency probe (< 5 MHz), either an abdominal or cardiac probe, positioned under the costal margin on the operated side and the contralateral side. To limit inter-operator variability, the patient's ultrasound evaluation will, as much as possible, be performed by the same operator. The presence of diaphragmatic dysfunction is defined by a diaphragmatic excursion of less than 1 cm.

SECONDARY OUTCOMES:
Pain evaluation | Hour 2
  Pain will be assessed using a simple numeric scale ranging from 0 (no pain) to 10 (worst pain ever experienced).
Pain evaluation | Hour 24
  Pain will be assessed using a simple numeric scale ranging from 0 (no pain) to 10 (worst pain ever experienced).
Diaphragmatic thickening evaluation | Hour 2
  Diaphragmatic thickening will be measured by ultrasound and will be assessed in relation to the baseline thickness and the contralateral diaphragmatic thickness
Diaphragmatic thickening evaluation | Hour 24
  Diaphragmatic thickening will be measured by ultrasound and will be assessed in relation to the baseline thickness and the contralateral diaphragmatic thickness
postoperative complications evaluation | Hour 2
  The screening for hypoxemia using a pulse oximeter will be conducted continuously throughout the study duration.
  Cardiovascular events will be evaluated based on the time to the occurrence of one of the 3 major cardiac events comprising the composite endpoint MACE (Major Adverse Cardiac Events): cardiovascular death, non-fatal myocardial infarction, non-fatal stroke.
postoperative complications evaluation | Hour 24
  The screening for hypoxemia using a pulse oximeter will be conducted continuously throughout the study duration.
  Cardiovascular events will be evaluated based on the time to the occurrence of one of the 3 major cardiac events comprising the composite endpoint MACE (Major Adverse Cardiac Events): cardiovascular death, non-fatal myocardial infarction, non-fatal stroke.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Claude Galien, Quincy-sous-Sénart, France

IPD SHARING:
Plan to Share IPD: Yes
Only data strictly relevant to and directly used in the published article will be eligible for sharing. No data outside the scope of the published analysis will be provided.
Supporting Information: ICF
Access Criteria: Data may be made available upon explicit request from the journal and solely for the purpose of conducting a re-analysis of the published results. Requests must be submitted by email to the corresponding author. The statistical code used for the original analyses may also be shared if necessary. The study authors may be invited to participate in the re-analysis depending on the nature of the request.
  Data will be provided as an anonymized Excel file, in compliance with applicable personal data protection regulations. No information allowing direct or indirect identification of study participants will be disclosed.
  Shared data may be used only for the purpose defined in the initial request. No secondary use, data transfer agreement, or further data exploitation will be authorized.

REFERENCES:
- [Derived] Guessous K, Elmaleh Y, Kattou F, Coblence M, Dore P, Zanoun N. Incidence of diaphragmatic dysfunction after non-intubated video-assisted thoracoscopic surgery: a prospective, single-centre observational study protocol. BMJ Open. 2025 Dec 31;15(12):e107479. doi: 10.1136/bmjopen-2025-107479. PMID 41475807